## 13.1 Anexo A: Hoja de información al paciente.



#### **IDENTIFICACIÓN DEL PACIENTE:**

## INTRODUCCIÓN

El investigador le ha explicado la posibilidad de participar en un estudio, sobre un nuevo manejo sin ingreso, tras la cirugía de apendicitis aguda no complicada

En este documento se le presenta la posibilidad que usted tiene de participar en un estudio experimental aleatorizado que consiste en comparar el manejo sin ingreso tras la intervención quirúrgica de apendicitis aguda no complicada. Ha de conocer que el presente estudio ha sido aprobado por el Comité Ético de Investigación Clínica correspondiente.

El investigador principal de este estudio es el Dr. Felipe Pareja Ciuro del la Unidad de Cirugía de Urgencias del hospital Universitario Virgen del Rocío.

La información que contiene este documento, que se conoce como Hoja de Información al Sujeto del ensayo, está destinada a que usted pueda conocer más a fondo este estudio y le ayude a decidir si quiere o no participar en el mismo.

Esta hoja de información puede contener palabras que usted no entienda. Por favor, pídale al investigador que desarrollará el estudio que le explique todas las palabras o la información que usted no comprenda claramente. Tómese el tiempo necesario para decidir si quiere o no participar en el presente estudio, consulte a personas de su confianza y pregunte cuanto sea necesario. Si decide no participar, esta decisión no afectará en modo alguno a su atención médica actual o futura.

#### **ANTECEDENTES**

Actualmente existen numerosas publicaciones sobre el manejo sin ingreso en pacientes con apendicitis aguda no complicada tras apendicectomía que señalan que puede ser seguro en pacientes seleccionados.

Este manejo pretende dar las ventajas de una cirugía sin ingreso, con brillantes resultados de actividad.

Entendemos como cirugía sin ingreso (CSI) como la atención a procesos quirúrgicos multidisciplinarios, realizados bajo cualquier tipo de anestesia y con unos cuidados postoperatorios poco intensivos, que permiten dar de alta al paciente a las pocas horas de finalizar el procedimiento. De acuerdo con esta definición inicial, el paciente vuelve a su domicilio el mismo día de la intervención y no requiere una cama hospitalaria. Se trata así de establecer diferencias con la cirugía menor ambulatoria, que engloba procedimientos quirúrgicos de muy baja complejidad realizados generalmente con anestesia local, y la cirugía de corta estancia, que hace referencia a procedimientos quirúrgicos que requieren una hospitalización de 1-2 días.

Por dicho motivo, se está investigando en este hospital la aplicabilidad de dicho manejo postquirúrgico para lo cual se ha planteado este estudio en el que tras realizarle la intervención quirúrgica usted podrá ser dado de alta desde la sala de reanimación postquirúrgica sin necesidad de ingreso en planta.

#### **OBJETIVOS DEL ESTUDIO**

El objetivo del estudio es evaluar la eficacia, seguridad y eficiencia de la cirugía sin ingreso en pacientes con apendicitis aguda no complicada a los que se les realiza una apendicectomía vía laparoscópica o abierta mediante incisión mínima. Se realizará un seguimiento durante un total de 1 mes +/- 30 días después de la finalización de la cirugía, con una revisión postoperatoria.

# ¿POR QUÉ SE LE HA PEDIDO QUE PARTICIPE?

Se le pide que participe porque usted ha sido diagnosticado de apendicitis aguda y hay que intervenirlo, de forma que tras la cirugía y si se encuentra bien, podrá ser dado de alta con los cuidados y consejos en domicilio que le facilitaremos.

El único modo de confirmar que régimen de alta es mejor es hacer dos grupos de pacientes de parecidas características y unos que se marchen con régimen de alta sin ingreso, mientras que los otros ingresarán planta de hospitalización. Para ello, usted será intervenido de igual forma sin cambios durante la técnica quirúrgica ni durante los cuidados postoperatorios.

## • <u>Visita 1 (Día-0)</u>:

Tras su admisión en urgencias por cuadro compatible con apendicitis aguda el paciente pasará a observación quirúrgica a cargo del Servicio de Cirugía General. Una vez ahí, se indicará la intervención quirúrgica, se realizará la selección de los pacientes y se informará del estudio a los pacientes seleccionados entregándoles el consentimiento informado para su participación. De igual forma para el grupo caso como para el grupo control.

Tras la pre-selección, los pacientes serán sometidos a apendicectomía tras la cual se realizará la inclusión definitiva (selección definitiva) y serán aleatorizados de manera ciega al grupo caso o al grupo control.

El paciente incluido en el grupo caso, será dado de alta en régimen de cirugía sin ingreso previo paso por la unidad de reanimación postanestésica donde será evaluada su correcta evolución postoperatoria así como su tolerancia a la dieta, micción espontanea, dolor controlado, entre otros.

En el caso del grupo control, el paciente ingresará en una planta de hospitalización a cargo de la Cirugía General y del Aparato Digestivo. El tiempo hasta el alta de estos pacientes estará determinado por el criterio del cirujano que lo intervino.

Previo al alta, el paciente rellenará la Escala de calidad de atención.

## • Visita 2 (1 mes +/- 30 días):

Revisión clínica, recogida de eventos adversos, y fin del estudio.

Si tiene alguna duda sobre las visitas del estudio y el tiempo que supondría para usted, no dude en preguntar al investigador responsable del desarrollo del estudio.

La visita de seguimiento del estudio se realizará de manera telefónica en horario laboral de lunes a viernes, en aproximadamente 1 mes +/- 30 días, por parte del investigador/es principal.

Si tiene alguna duda sobre la visita evolutiva y el tiempo que supondría para usted, no dude en preguntar al investigador responsable del desarrollo del estudio.

La visita mencionada se realizará de manera telefónica, en día laboral

## **DURACIÓN DEL ESTUDIO**

Su participación en el estudio tendrá una duración de 1 mes +/- 30 días, durante el mismo usted recibirá una consulta telefónica por parte del investigador/es del estudio que permitirán controlar la evolución de su enfermedad, momento en que se finalizará el estudio.

Según el protocolo de este estudio, se estima que el mismo dure 24 meses: 18 meses de reclutamiento, un periodo de 1 mes +/- 30 días de seguimiento y finalmente 4 meses de análisis de los datos.

#### **BENEFICIOS ESPERADOS**

Existe la posibilidad de que, al tratarse de un manejo postoperatorio que se encuentra actualmente en investigación usted no obtenga un beneficio directo por su participación en el estudio, ya que éste es uno de los aspectos que se pretende llegar a conocer con la realización del mismo. En este supuesto, con su participación en el estudio, usted habrá contribuido a tener un mejor conocimiento de su enfermedad y a que se puedan continuar estudiando nuevas posibilidades de tratamiento.

## RIESGOS DERIVADOS DE SU PARTICIPACIÓN EN EL ESTUDIO

El riesgo de complicaciones es bajo. No obstante, debe saber que no está exento de los riesgos inherentes a cualquier tratamiento propio de la cirugía y no derivado del estudio, explicados ya en su consentimiento informado pertinente. La aparición de las referidas complicaciones dependerá de la circunstancia basal de cada sujeto, a su vez.

En caso de no querer participar en el estudio que se le propone, el investigador responsable le indicará las alternativas actualmente disponibles, que en este caso será el ingreso a planta.

No dude en consultar con el investigador responsable del desarrollo del estudio cualquier duda que tenga por este motivo.

Alergias manifestadas por el paciente:

Si usted tiene alergia a algún medicamento, asma u otras enfermedades alérgicas, si padece del corazón o tiene una insuficiencia renal, debe ponerlo en conocimiento del personal facultativo encargado de la prueba.

Riesgos graves e infrecuentes:

Hasta el momento no se han descrito efectos graves con el manejo sin ingreso a estudio.

# CARÁCTER VOLUNTARIO DE LA PARTICIPACIÓN Y POSIBILIDAD DE RETIRARSE DEL ESTUDIO

Su participación en este estudio es voluntaria y puede abandonarlo en cualquier momento si lo desea, sin tener que dar explicación alguna, bastando simplemente con firmar el recuadro de revocación del consentimiento prestado para la participación en el estudio.

Si usted abandona voluntariamente el estudio o algún médico le pide que lo haga, deberá notificárselo al investigador. Ni su asistencia médica habitual ni la relación con el investigador se verá afectada por dejar de participar en el estudio. En dicho caso, es conveniente que siga las indicaciones del investigador para proceder de la mejor manera a la finalización ordenada de las actividades derivadas de su participación en estudio, es decir, realizando las actividades propias de la última visita o visita final.

También debe saber que, el estudio o su participación en el mismo podrían terminar en cualquier momento, sin que sea necesario obtener su consentimiento, por razones médicas o circunstancias no previsibles, siempre que el promotor, investigador o autoridades sanitarias lo consideren oportuno.

El investigador que desarrolla el estudio puede decidir suspender su participación en el mismo, si considera que es lo mejor para usted o en caso de que usted no siga los procedimientos del ensayo. Asimismo, él le informará de cualquier hallazgo significativo, que pueda estar relacionado con su participación.

## **CONTRAINDICACIONES**

Se considerarán criterios de exclusión de los pacientes previamente seleccionados, los que se enumeran a continuación:

- Hallazgos intraoperatorios que sugieran: Absceso o plastrón apendicular, Peritonitis focalizada o difusa, Apendicitis aguda complicada: apendicitis gangrenosa, perforada, con absceso o con abundante líquido libre intraabdominal
- Necesidad de colocación de drenaje abdominal.
- Dudas en el diagnóstico definitivo.
- Sospecha de enfermedad inflamatoria intestinal.
- No soporte familiar.
- No firma de consentimiento informado.
- Imposibilidad del cumplimento del seguimiento.

# CONFIDENCIALIDAD DE DATOS PERSONALES Y ACCESO A LA HISTORIA CLÍNICA DEL PACIENTE

El tratamiento, la comunicación y la cesión de los datos de carácter personal de todos los sujetos participantes en el estudio se ajustarán a lo dispuesto en la Ley Orgánica 15/1999, de 13 de diciembre, de Protección de Datos de Carácter Personal.

Usted podrá ejercitar los derechos reconocidos a los interesados en la citada Ley Orgánica, es decir, los derechos de acceso, rectificación, oposición y cancelación de sus datos personales, con las limitaciones establecidas en dicha Ley Orgánica. Para ello, deberá dirigirse al investigador. Asimismo, debe usted saber que su historia clínica será guardada por imperativo de la Ley 41/2002, de 14 de noviembre, básica reguladora de la autonomía del paciente y de derechos y obligaciones en materia de documentación e información clínica, durante al menos cinco años a contar desde el último episodio asistencial.

Al firmar el consentimiento informado usted autoriza a un representante del promotor o del Comité Ético de Investigación Clínica de su hospital, para el acceso a su historia clínica con la finalidad de verificar las informaciones clínicas, que se vayan generando durante el estudio, así como el acceso a sus datos personales y datos clínicos, y la cesión de estos única y exclusivamente con la finalidad para la que fueron recabados.

Sólo tendrá acceso a su información personal e historia clínica el personal autorizado para ello, esto es, el investigador principal y equipo de investigación, las autoridades sanitarias, los Comités Éticos de Investigación Clínica y el personal autorizado por el promotor, cuando lo precisen para comprobar los datos y procedimientos del estudio, pero siempre manteniendo la confidencialidad de los mismos de acuerdo a la legislación vigente. Sus datos clínicos pueden ser

transferidos a otras empresas que trabajen en representación del promotor en este programa de investigación, incluso a empresas fuera del área económica europea (AEE).

No obstante lo anterior, el responsable del estudio garantizará en todo momento la confidencialidad de sus datos personales y datos clínicos, y actuará en todo momento conforme a lo establecido en la Ley Orgánica 15/1999, de 13 de diciembre, de Protección de Datos de Carácter Personal.

Los registros del estudio que se obtengan con el fin de analizar los resultados se identificarán únicamente con un número que le será asignado en el momento de su inclusión en el estudio, para evitar revelar su identidad fuera del hospital y sólo el investigador y sus colaboradores podrán relacionar tales datos con usted y su historia clínica. Por dicho motivo, su identidad no será revelada a persona alguna salvo excepciones, en caso de urgencia médica o requerimiento legal.

No obstante lo anterior, sólo se transmitirán al promotor los datos personales necesarios para cubrir el objetivo de dicho ensayo. Además, únicamente se accederá a la parte de la historia clínica cuyos datos sean relevantes para el estudio, y en cualquier caso, siempre se guardará la más estricta confidencialidad.

Su identidad no será revelada en ningún momento durante el estudio y, si sus datos se analizan y anotan en un informe, cuando los resultados de este ensayo se publiquen, se garantiza que su identidad permanecerá oculta.

## **RESPONSABILIDADES DEL PACIENTE**

Como paciente que participa voluntariamente en este estudio, tiene la responsabilidad de acudir a todas las visitas programadas del mismo, informar en la visita al investigador de todo lo que le haya ocurrido, de todos los medicamentos que esté tomando y de todos los sucesos secundarios que pudiera experimentar.

## COSTES POR SU PARTICIPACIÓN EN EL ESTUDIO

Su participación en el estudio, el tratamiento que reciba o los procedimientos que se requieran no le ocasionarán a usted gasto alguno.

## ASPECTOS ÉTICOS DEL ESTUDIO

El estudio se llevará a cabo de acuerdo a Normas de Buena Práctica Clínica (ICH-GCP), los principios contenidos en la declaración de Helsinki, el Convenio de Oviedo y la legislación española en materia de ensayos clínicos (Real Decreto 223/2004).

PREGUNTAS E INFORMACIÓN: PERSONAS DE CONTACTO

Usted puede realizar cuantas preguntas considere oportunas antes de otorgar su consentimiento informado por escrito. Cualquier nueva información referente al tratamiento que reciba y que se descubra durante su participación, le será debidamente comunicada y se le dará la oportunidad, si así lo desea, de revocar su consentimiento informado para la participación en el estudio.

Usted puede realizar todas las preguntas que desee y saber más sobre este estudio ahora o en cualquier momento en el curso del mismo. Además, si experimenta cualquier reacción adversa, debe contactar inmediatamente con el investigador, para ello podrá contactar con:

Dr.: Tallón Aguilar o Durán Muñoz Teléfono: 695956555 / 695956520

Usted tiene que decidir si participa o no. Si decide participar se le proporcionará esta hoja de información, donde deberá firmar el consentimiento informado para su participación. A usted se le entregará una copia de este documento y el investigador responsable del desarrollo del estudio se quedará con el documento original.

Si decide participar, es libre de revocar su consentimiento informado en cualquier momento y sin tener que dar explicaciones. Ello no afectará a la calidad de la atención que usted reciba. Si decide retirarse del estudio, el investigador le comentará la mejor forma de terminar dicho ensayo de forma ordenada.

# 13.2 Anexo B: Consentimiento informado.

Título del proyecto: " ENSAYO CLÍNICO UNICÉNTRICO, ALEATORIZADO, DOBLE CIEGO, PARA EVALUAR LA SEGURIDAD Y LA EFICACIA DEL ALTA EN RÉGIMEN DE CIRUGÍA SIN INGRESO EN PACIENTES CON APENDICITIS AGUDA INTERVENIDOS DE URGENCIAS".

| Investigador Principal: Dr. Felipe Pareja (<br>Hospital Universitario Virgen del Rocío de Se | _ |
|---|---|
| Yo,el Dr. investigación arriba mencionado, y declaro c | , colaborador del proyecto de |
| He leído la Hoja de Información que se me h | a entregado. |
| He podido hacer preguntas sobre el estudio. | |
| He recibido respuesta satisfactorias a mis preguntas. | |
| He recibido suficiente información sobre el estudio. | |
| Comprendo que mi participación es voluntaria | |
| Comprendo que todos mis datos serán tratados confidencialmente. | |
| Comprendo que puedo retirarme del estudio cuando quiera sin tener que dar explicaciones. Sin que esto repercuta en mis cuidados médicos. | |
| Mediante este acto Vd. consiente el uso de sus muestras en relación con este proyecto de investigación. SiNo | |
| Doy mi conformidad para participar en este estudio, | |
| Firma del paciente: | Firma del Investigador: |
| Fecha | Fecha |